CLINICAL TRIAL: NCT06931574
Title: Comparison of Cardiovascular Outcomes of Double Kissing-crush vs Controlled Balloon-crush Techniques For Complex Coronary Bifurcation Lesions
Brief Title: Double Kissing-crush vs Controlled Balloon-crush Techniques For Complex Coronary Bfurcation Lesions
Status: Recruiting | Type: Observational
Sponsor: Istanbul Mehmet Akif Ersoy Educational and Training Hospital (Other Government)
Collaborators: Sisli Hamidiye Etfal Training and Research Hospital (Other); Başakşehir Çam & Sakura City Hospital (Other Government); Bagcilar Training and Research Hospital (Other Government); Ankara Etlik City Hospital (Other Government); Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government); Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital (Other); Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Ahmet Guner, Principal Investigator, Istanbul Mehmet Akif Ersoy Educational and Training Hospital
Other Study IDs: 2025.03-21
Record Dates: First submitted 2025-04-08; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Coronary Arterial Disease (CAD); Percutaneous Coronary Intervention (PCI); Bifurcation Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Controlled balloon-crush Group
- Double kissing-crush stenting Group

SUMMARY:
The Crush technique for coronary bifurcation lesions has evolved significantly since its introduction to the literature by Colombo et al. in 2003, with several iterations, including double kissing balloon inflation. The main disadvantage of the historical Crush technique is the low success rate of the final kissing balloon inflation. An improvement came with the introduction of double kissing crush stenting aiming for the shorter protrusion and kissing balloon dilation performed before and after main branch stent implantation. The double kissing crush provides a significant reduction in major adverse cardiovascular events compared to Provisional stenting, Crush, and Culotte techniques. Recently, a novel modified mini-crush technique (controlled balloon-crush) has been introduced to the literature and is one of the most up-to-date crush techniques. The main advantage of this technique over the contemporary mini-crush technique is that the side branch can be easily rewired, and the 1:1 size non-compliant balloon can easily pass through the crushed stent structure in the ostial part of the side branch. The basic rationale of this is that the crushing of the side branch stent is done in a more controlled manner (by slowly deflation of the side branch stent balloon), and this causes less disruption of the stent cells. To date, no data compares the mid-term outcomes of double kissing crush and controlled balloon-crush stenting techniques in patients with complex coronary bifurcation lesions. Hence, this study aimed to determine the clinical results of double kissing crush and controlled balloon-crush techniques under mid-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18
* PCI with either DK-crush or Controlled balloon-crush
* Complex coronary bifurcation lesion (Medina 0.1.1, Medina 1.1.1)

Exclusion Criteria:

* Non-complex bifurcation anatomy
* Bail-out 2-stent (reverse modified mini-crush)
* ST-elevation myocardial infarction
* Cardiogenic shock status
* In-stent restenosis
* A previous of coronary artery bypass grafting
* Implantation of bare-metal stent
* End-stage hepatic or renal disease
* <1-year life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Complex coronary bifurcation disease
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint (Target lesion failure) | 36 months
  Target lesion failure (%) is defined as the combination of cardiac death (%), target vessel myocardial infarction (%), or target lesion revascularization (%) rates.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Mehmet Akif Ersoy Thoracic and Cardiovascular Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided